CLINICAL TRIAL: NCT05746299
Title: The Emergence of Abstract Structure Knowledge Across Learning and Sleep
Brief Title: The Impact of Reactivation During Sleep on the Consolidation of Abstract Information in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 833228A; 1R21MH128788-01A1 (NIH)
Record Dates: First submitted 2023-02-14; First posted 2023-02-27 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Memory Consolidation
Keywords: memory; sleep; learning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Immediate Congruent (Experimental): Participants will learn and be tested on two different semantic categories with the same structure that dictates the co-occurrence of different features.
  Interventions: Behavioral: Congruent vs. Incongruent; Behavioral: Immediate vs. Awake vs. Asleep
- Immediate Incongruent (Experimental): Participants will learn and be tested on two different semantic categories with different structures that dictate the co-occurrence of different features.
  Interventions: Behavioral: Congruent vs. Incongruent; Behavioral: Immediate vs. Awake vs. Asleep
- Awake Incongruent (Experimental): Participants will learn two different semantic categories, neither of which has a Modular structure. After a 2.5-hour break, they will learn and be tested on a novel semantic category with a Modular structure.
  Interventions: Behavioral: Congruent vs. Incongruent; Behavioral: Immediate vs. Awake vs. Asleep
- Awake Congruent (Experimental): Participants will learn two different semantic categories, one of which has a Modular structure. After a 2.5-hour break, they will learn and be tested on a novel semantic category with a Modular structure.
  Interventions: Behavioral: Congruent vs. Incongruent; Behavioral: Immediate vs. Awake vs. Asleep
- Sleep Incongruent (Experimental): Participants will learn two different semantic categories, one of which has a Modular structure. After a 2-hour nap opportunity, during which TMR will be used to reactivate the non-Modular category, participants will take a 30-minute break. After the break, they will learn and be tested on a novel semantic category with a Modular structure.
  Interventions: Behavioral: Congruent vs. Incongruent; Behavioral: Immediate vs. Awake vs. Asleep; Behavioral: Targeted memory reactivation (TMR)
- Sleep Congruent (SWS) (Experimental): Participants will learn two different semantic categories, one of which has a Modular structure. After a 2-hour nap opportunity, during which TMR will be used to reactivate the Modular category during slow wave sleep (SWS), participants will take a 30-minute break. After the break, they will learn and be tested on a novel semantic category with a Modular structure.
  Interventions: Behavioral: Congruent vs. Incongruent; Behavioral: Immediate vs. Awake vs. Asleep; Behavioral: Targeted memory reactivation (TMR)
- Sleep Congruent (REM) (Experimental): Participants will learn two different semantic categories, one of which has a Modular structure. After a 2-hour nap opportunity, during which TMR will be used to reactivate the Modular category during rapid eye movement (REM) sleep, participants will take a 30-minute break. After the break, they will learn and be tested on a novel semantic category with a Modular structure.
  Interventions: Behavioral: Congruent vs. Incongruent; Behavioral: Immediate vs. Awake vs. Asleep; Behavioral: Targeted memory reactivation (TMR)

INTERVENTIONS:
Behavioral: Congruent vs. Incongruent — The Congruent vs. Incongruent intervention relates to the feature-based structure of the novel categories (Modular or non-Modular) and whether there is (Congruent) or is not (Incongruent) a match between what was previously learned and the final target category.
Behavioral: Immediate vs. Awake vs. Asleep — Immediate, Awake, and Sleep refer to either no break, 2.5 hours awake, or 2 hours asleep plus a 30-minute post-nap break to account for sleep inertia between learning and target category.
Behavioral: Targeted memory reactivation (TMR) — Targeted memory reactivation (TMR) is the systematic presentation of sounds during sleep that were associated with certain stimuli during learning and will be administered either during slow wave sleep (SWS) or rapid eye movement (REM) sleep.
  Arms: Sleep Congruent (REM); Sleep Congruent (SWS); Sleep Incongruent

SUMMARY:
In any given cognitive domain, representations of individual elements are not independent but are organized by means of structured relations. Representations of this underlying structure are powerful, allowing generalization and inference in novel environments. In the semantic domain, structure captures associations between different semantic features or concepts (e.g., green, wings, can fly) and is known to influence the development and deterioration of semantic knowledge. The investigators recently found that humans more easily learn novel categories that contain clusters of reliably co-occurring features, revealing an influence of structure on novel category formation. However, a critical unknown is whether learned representations of structure are closely tied to category-specific elements, or whether such representations become abstract to some extent, transformed away from the experienced features. Further, if abstract structural representations do emerge, prior work provides intriguing hints that these representations may require offline consolidation during awake rest or sleep. The investigators have developed a paradigm in which carefully designed graph structures govern the pattern of feature co-occurrences within individual categories. Here the investigators implement a "structure transfer" extension of this paradigm in order to determine whether learning one structured category facilitates learning of a second identically structured category defined by a new set of features. This facilitation would provide evidence that structure representations are abstract to some degree. Aim 1 will use these methods to evaluate whether abstract structural representations emerge immediately during learning. Aim 2 will determine whether these representations persist, or emerge, over a delay, and whether sleep-based consolidation in particular is needed. The role of replay of recent experience during sleep will be evaluated using electroencephalography (EEG) paired with closed-loop targeted memory reactivation (TMR), a technique that enables causal influence over the consolidation of recently learned information in humans. This work will inform and constrain theories of semantic learning as well as theories of structure learning and representation more broadly.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18 and 35

Exclusion Criteria:

* No medical or neurological illness that would impact experimental performance
* Not a member of a vulnerable population

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 194 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna C Schapiro, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Time Frame: IPD will be available at the time of study publication.
Access Criteria: IPD will be publicly available without restriction.

REFERENCES:
- [Background] Gentner, D.. Structure-mapping: A theoretical framework for analogy. Cognitive science. 1983;7(2): 155-170.
- [Background] Thibodeau PH, Flusberg SJ, Glick JJ, & Sternberg DA. An emergent approach to analogical inference. Connection Science. 2013; 25(1): 27-53.
- [Background] Collins AGE, Frank MJ. Neural signature of hierarchically structured expectations predicts clustering and transfer of rule sets in reinforcement learning. Cognition. 2016 Jul;152:160-169. doi: 10.1016/j.cognition.2016.04.002. Epub 2016 Apr 12. PMID 27082659
- [Background] Baram AB, Muller TH, Nili H, Garvert MM, Behrens TEJ. Entorhinal and ventromedial prefrontal cortices abstract and generalize the structure of reinforcement learning problems. Neuron. 2021 Feb 17;109(4):713-723.e7. doi: 10.1016/j.neuron.2020.11.024. Epub 2020 Dec 22. PMID 33357385
- [Background] TOLMAN EC. Cognitive maps in rats and men. Psychol Rev. 1948 Jul;55(4):189-208. doi: 10.1037/h0061626. No abstract available. PMID 18870876
- [Background] Behrens TEJ, Muller TH, Whittington JCR, Mark S, Baram AB, Stachenfeld KL, Kurth-Nelson Z. What Is a Cognitive Map? Organizing Knowledge for Flexible Behavior. Neuron. 2018 Oct 24;100(2):490-509. doi: 10.1016/j.neuron.2018.10.002. PMID 30359611
- [Background] Whittington JCR, Muller TH, Mark S, Chen G, Barry C, Burgess N, Behrens TEJ. The Tolman-Eichenbaum Machine: Unifying Space and Relational Memory through Generalization in the Hippocampal Formation. Cell. 2020 Nov 25;183(5):1249-1263.e23. doi: 10.1016/j.cell.2020.10.024. Epub 2020 Nov 11. PMID 33181068
- [Background] McClelland JL, Rogers TT. The parallel distributed processing approach to semantic cognition. Nat Rev Neurosci. 2003 Apr;4(4):310-22. doi: 10.1038/nrn1076. No abstract available. PMID 12671647
- [Background] Solomon SH, Schapiro AC. Structure shapes the representation of a novel category. J Exp Psychol Learn Mem Cogn. 2024 Mar;50(3):458-483. doi: 10.1037/xlm0001257. Epub 2023 Jun 15. PMID 37326540
- [Background] Bahdanau D, Murty S, Noukhovitch M, Nguyen TH, de Vries H, Courville A. Systematic generalization: what is required and can it be learned?. arXiv preprint. 2018.
- [Background] Mark S, Moran R, Parr T, Kennerley SW, Behrens TEJ. Transferring structural knowledge across cognitive maps in humans and models. Nat Commun. 2020 Sep 22;11(1):4783. doi: 10.1038/s41467-020-18254-6. PMID 32963219
- [Background] Durrant SJ, Cairney SA, Lewis PA. Cross-modal transfer of statistical information benefits from sleep. Cortex. 2016 May;78:85-99. doi: 10.1016/j.cortex.2016.02.011. Epub 2016 Feb 27. PMID 27017231
- [Background] Tamminen J, Lambon Ralph MA, Lewis PA. Targeted memory reactivation of newly learned words during sleep triggers REM-mediated integration of new memories and existing knowledge. Neurobiol Learn Mem. 2017 Jan;137:77-82. doi: 10.1016/j.nlm.2016.11.012. Epub 2016 Nov 15. PMID 27864086
- [Background] Wang B, Antony JW, Lurie S, Brooks PP, Paller KA, Norman KA. Targeted Memory Reactivation during Sleep Elicits Neural Signals Related to Learning Content. J Neurosci. 2019 Aug 21;39(34):6728-6736. doi: 10.1523/JNEUROSCI.2798-18.2019. Epub 2019 Jun 24. PMID 31235649
- [Background] Schapiro AC, Turk-Browne NB, Norman KA, Botvinick MM. Statistical learning of temporal community structure in the hippocampus. Hippocampus. 2016 Jan;26(1):3-8. doi: 10.1002/hipo.22523. Epub 2015 Oct 13. PMID 26332666
- [Background] Mack ML, Love BC, Preston AR. Building concepts one episode at a time: The hippocampus and concept formation. Neurosci Lett. 2018 Jul 27;680:31-38. doi: 10.1016/j.neulet.2017.07.061. Epub 2017 Aug 8. PMID 28801273
- [Background] Weickert TW, Goldberg TE, Callicott JH, Chen Q, Apud JA, Das S, Zoltick BJ, Egan MF, Meeter M, Myers C, Gluck MA, Weinberger DR, Mattay VS. Neural correlates of probabilistic category learning in patients with schizophrenia. J Neurosci. 2009 Jan 28;29(4):1244-54. doi: 10.1523/JNEUROSCI.4341-08.2009. PMID 19176832
- [Background] Monti JM, Monti D. Sleep disturbance in schizophrenia. Int Rev Psychiatry. 2005 Aug;17(4):247-53. doi: 10.1080/09540260500104516. PMID 16194796
- [Background] Tsuno N, Besset A, Ritchie K. Sleep and depression. J Clin Psychiatry. 2005 Oct;66(10):1254-69. doi: 10.4088/jcp.v66n1008. PMID 16259539
- [Background] Riemann D, Berger M, Voderholzer U. Sleep and depression--results from psychobiological studies: an overview. Biol Psychol. 2001 Jul-Aug;57(1-3):67-103. doi: 10.1016/s0301-0511(01)00090-4. PMID 11454435
- [Background] Nutt D, Wilson S, Paterson L. Sleep disorders as core symptoms of depression. Dialogues Clin Neurosci. 2008;10(3):329-36. doi: 10.31887/DCNS.2008.10.3/dnutt. PMID 18979946
- [Background] Karuza EA, Kahn AE, Bassett DS. Human sensitivity to community structure is robust to topological variation. Complexity. 2019.
- [Background] Karuza EA, Kahn AE, Thompson-Schill SL, Bassett DS. Process reveals structure: How a network is traversed mediates expectations about its architecture. Sci Rep. 2017 Oct 6;7(1):12733. doi: 10.1038/s41598-017-12876-5. PMID 28986524
- [Background] Karuza EA, Thompson-Schill SL, Bassett DS. Local Patterns to Global Architectures: Influences of Network Topology on Human Learning. Trends Cogn Sci. 2016 Aug;20(8):629-640. doi: 10.1016/j.tics.2016.06.003. Epub 2016 Jun 29. PMID 27373349
- [Background] Lynn CW, Bassett DS. How humans learn and represent networks. Proc Natl Acad Sci U S A. 2020 Nov 24;117(47):29407-29415. doi: 10.1073/pnas.1912328117. PMID 33229528
- [Background] Schapiro AC, Rogers TT, Cordova NI, Turk-Browne NB, Botvinick MM. Neural representations of events arise from temporal community structure. Nat Neurosci. 2013 Apr;16(4):486-92. doi: 10.1038/nn.3331. Epub 2013 Feb 17. PMID 23416451
- [Background] Kahn AE, Karuza EA, Vettel JM, Bassett DS. Network constraints on learnability of probabilistic motor sequences. Nat Hum Behav. 2018 Dec;2(12):936-947. doi: 10.1038/s41562-018-0463-8. Epub 2018 Nov 5. PMID 30988437
- [Background] Kakaei E, Aleshin S, Braun J. Visual object recognition is facilitated by temporal community structure. Learn Mem. 2021 Apr 15;28(5):148-152. doi: 10.1101/lm.053306.120. Print 2021 May. PMID 33858967
- [Background] Eichenbaum H. Time cells in the hippocampus: a new dimension for mapping memories. Nat Rev Neurosci. 2014 Nov;15(11):732-44. doi: 10.1038/nrn3827. Epub 2014 Oct 1. PMID 25269553
- [Background] Moser MB, Rowland DC, Moser EI. Place cells, grid cells, and memory. Cold Spring Harb Perspect Biol. 2015 Feb 2;7(2):a021808. doi: 10.1101/cshperspect.a021808. PMID 25646382
- [Background] Maguire EA, Spiers HJ, Good CD, Hartley T, Frackowiak RS, Burgess N. Navigation expertise and the human hippocampus: a structural brain imaging analysis. Hippocampus. 2003;13(2):250-9. doi: 10.1002/hipo.10087. PMID 12699332
- [Background] Kumaran D, McClelland JL. Generalization through the recurrent interaction of episodic memories: a model of the hippocampal system. Psychol Rev. 2012 Jul;119(3):573-616. doi: 10.1037/a0028681. PMID 22775499
- [Background] Cohen N., Eichenbaum H. Memory, amnesia, and the hippocampal system. MIT press. 1993.
- [Background] Belal S, Cousins J, El-Deredy W, Parkes L, Schneider J, Tsujimura H, Zoumpoulaki A, Perapoch M, Santamaria L, Lewis P. Identification of memory reactivation during sleep by EEG classification. Neuroimage. 2018 Aug 1;176:203-214. doi: 10.1016/j.neuroimage.2018.04.029. Epub 2018 Apr 17. PMID 29678758
- [Background] Stickgold R. Sleep-dependent memory consolidation. Nature. 2005 Oct 27;437(7063):1272-8. doi: 10.1038/nature04286. PMID 16251952
- [Background] Rasch B, Born J. About sleep's role in memory. Physiol Rev. 2013 Apr;93(2):681-766. doi: 10.1152/physrev.00032.2012. PMID 23589831
- [Background] Wagner U, Gais S, Haider H, Verleger R, Born J. Sleep inspires insight. Nature. 2004 Jan 22;427(6972):352-5. doi: 10.1038/nature02223. PMID 14737168
- [Background] Ellenbogen JM, Hu PT, Payne JD, Titone D, Walker MP. Human relational memory requires time and sleep. Proc Natl Acad Sci U S A. 2007 May 1;104(18):7723-8. doi: 10.1073/pnas.0700094104. Epub 2007 Apr 20. PMID 17449637
- [Background] Schapiro AC, McDevitt EA, Chen L, Norman KA, Mednick SC, Rogers TT. Sleep Benefits Memory for Semantic Category Structure While Preserving Exemplar-Specific Information. Sci Rep. 2017 Nov 1;7(1):14869. doi: 10.1038/s41598-017-12884-5. PMID 29093451
- [Background] Lewis PA, Knoblich G, Poe G. How Memory Replay in Sleep Boosts Creative Problem-Solving. Trends Cogn Sci. 2018 Jun;22(6):491-503. doi: 10.1016/j.tics.2018.03.009. PMID 29776467
- [Background] Feld GB, Bernard M, Rawson AB, Spiers HJ. Sleep targets highly connected global and local nodes to aid consolidation of learned graph networks. Sci Rep. 2022 Sep 5;12(1):15086. doi: 10.1038/s41598-022-17747-2. PMID 36064730
- [Background] McClelland JL, McNaughton BL, O'Reilly RC. Why there are complementary learning systems in the hippocampus and neocortex: insights from the successes and failures of connectionist models of learning and memory. Psychol Rev. 1995 Jul;102(3):419-457. doi: 10.1037/0033-295X.102.3.419. PMID 7624455
- [Background] Marshall L, Born J. The contribution of sleep to hippocampus-dependent memory consolidation. Trends Cogn Sci. 2007 Oct;11(10):442-50. doi: 10.1016/j.tics.2007.09.001. Epub 2007 Oct 1. PMID 17905642
- [Background] Davidson TJ, Kloosterman F, Wilson MA. Hippocampal replay of extended experience. Neuron. 2009 Aug 27;63(4):497-507. doi: 10.1016/j.neuron.2009.07.027. PMID 19709631
- [Background] Schapiro AC, McDevitt EA, Rogers TT, Mednick SC, Norman KA. Human hippocampal replay during rest prioritizes weakly learned information and predicts memory performance. Nat Commun. 2018 Sep 25;9(1):3920. doi: 10.1038/s41467-018-06213-1. PMID 30254219
- [Background] Cairney SA, Durrant SJ, Hulleman J, Lewis PA. Targeted memory reactivation during slow wave sleep facilitates emotional memory consolidation. Sleep. 2014 Apr 1;37(4):701-7, 707A. doi: 10.5665/sleep.3572. PMID 24688163
- [Background] Batterink LJ, Paller KA. Sleep-based memory processing facilitates grammatical generalization: Evidence from targeted memory reactivation. Brain Lang. 2017 Apr;167:83-93. doi: 10.1016/j.bandl.2015.09.003. Epub 2015 Oct 9. PMID 26443322
- [Background] Goldi M, van Poppel EAM, Rasch B, Schreiner T. Increased neuronal signatures of targeted memory reactivation during slow-wave up states. Sci Rep. 2019 Feb 25;9(1):2715. doi: 10.1038/s41598-019-39178-2. PMID 30804371
- [Background] Ngo HV, Martinetz T, Born J, Molle M. Auditory closed-loop stimulation of the sleep slow oscillation enhances memory. Neuron. 2013 May 8;78(3):545-53. doi: 10.1016/j.neuron.2013.03.006. Epub 2013 Apr 11. PMID 23583623
- [Background] Ngo HV, Miedema A, Faude I, Martinetz T, Molle M, Born J. Driving sleep slow oscillations by auditory closed-loop stimulation-a self-limiting process. J Neurosci. 2015 Apr 29;35(17):6630-8. doi: 10.1523/JNEUROSCI.3133-14.2015. PMID 25926443
- [Background] Navarrete M, Schneider J, Ngo HV, Valderrama M, Casson AJ, Lewis PA. Examining the optimal timing for closed-loop auditory stimulation of slow-wave sleep in young and older adults. Sleep. 2020 Jun 15;43(6):zsz315. doi: 10.1093/sleep/zsz315. PMID 31872860
- [Background] Solomon SH, Medaglia JD, Thompson-Schill SL. Implementing a concept network model. Behav Res Methods. 2019 Aug;51(4):1717-1736. doi: 10.3758/s13428-019-01217-1. PMID 30891712
- [Background] Collins AM, Loftus EF. A spreading-activation theory of semantic processing. Psychological review. 1975; 82(6): 407.
- [Background] De Deyne S, Navarro DJ, Perfors A, Storms G. Structure at every scale: A semantic network account of the similarities between unrelated concepts. J Exp Psychol Gen. 2016 Sep;145(9):1228-54. doi: 10.1037/xge0000192. PMID 27560855
- [Background] McRae K, de Sa VR, Seidenberg MS. On the nature and scope of featural representations of word meaning. J Exp Psychol Gen. 1997 Jun;126(2):99-130. doi: 10.1037//0096-3445.126.2.99. PMID 9163932
- [Background] Tyler LK, Moss HE, Durrant-Peatfield MR, Levy JP. Conceptual structure and the structure of concepts: a distributed account of category-specific deficits. Brain Lang. 2000 Nov;75(2):195-231. doi: 10.1006/brln.2000.2353. PMID 11049666
- [Background] Saffran JR, Johnson EK, Aslin RN, Newport EL. Statistical learning of tone sequences by human infants and adults. Cognition. 1999 Feb 1;70(1):27-52. doi: 10.1016/s0010-0277(98)00075-4. PMID 10193055
- [Background] Saffran JR. The use of predictive dependencies in language learning. Journal of Memory and Language. 2001; 44(4): 493-515.
- [Background] Fiser J, Aslin RN. Statistical learning of new visual feature combinations by infants. Proc Natl Acad Sci U S A. 2002 Nov 26;99(24):15822-6. doi: 10.1073/pnas.232472899. Epub 2002 Nov 12. PMID 12429858
- [Background] Kirkham NZ, Slemmer JA, Johnson SP. Visual statistical learning in infancy: evidence for a domain general learning mechanism. Cognition. 2002 Mar;83(2):B35-42. doi: 10.1016/s0010-0277(02)00004-5. PMID 11869728
- [Background] Pearce MT, Ruiz MH, Kapasi S, Wiggins GA, Bhattacharya J. Unsupervised statistical learning underpins computational, behavioural, and neural manifestations of musical expectation. Neuroimage. 2010 Mar;50(1):302-13. doi: 10.1016/j.neuroimage.2009.12.019. Epub 2009 Dec 11. PMID 20005297
- [Background] Turk-Browne NB, Junge J, Scholl BJ. The automaticity of visual statistical learning. J Exp Psychol Gen. 2005 Nov;134(4):552-64. doi: 10.1037/0096-3445.134.4.552. PMID 16316291
- [Background] O'Keefe J, Nadel L. The hippocampus as a cognitive map. Oxford university press. 1978.
- [Background] Hafting T, Fyhn M, Molden S, Moser MB, Moser EI. Microstructure of a spatial map in the entorhinal cortex. Nature. 2005 Aug 11;436(7052):801-6. doi: 10.1038/nature03721. Epub 2005 Jun 19. PMID 15965463
- [Background] Javadi AH, Emo B, Howard LR, Zisch FE, Yu Y, Knight R, Pinelo Silva J, Spiers HJ. Hippocampal and prefrontal processing of network topology to simulate the future. Nat Commun. 2017 Mar 21;8:14652. doi: 10.1038/ncomms14652. PMID 28323817
- [Background] Killian NJ, Buffalo EA. Grid cells map the visual world. Nat Neurosci. 2018 Feb;21(2):161-162. doi: 10.1038/s41593-017-0062-4. No abstract available. PMID 29371658
- [Background] Stachenfeld KL, Botvinick MM, Gershman SJ. The hippocampus as a predictive map. Nat Neurosci. 2017 Nov;20(11):1643-1653. doi: 10.1038/nn.4650. Epub 2017 Oct 2. PMID 28967910
- [Background] Epstein RA, Patai EZ, Julian JB, Spiers HJ. The cognitive map in humans: spatial navigation and beyond. Nat Neurosci. 2017 Oct 26;20(11):1504-1513. doi: 10.1038/nn.4656. PMID 29073650
- [Background] Erickson JE, Chin-Parker S, Ross BH. Inference and classification learning of abstract coherent categories. J Exp Psychol Learn Mem Cogn. 2005 Jan;31(1):86-99. doi: 10.1037/0278-7393.31.1.86. PMID 15641907
- [Background] Park SA, Miller DS, Boorman ED. Inferences on a multidimensional social hierarchy use a grid-like code. Nat Neurosci. 2021 Sep;24(9):1292-1301. doi: 10.1038/s41593-021-00916-3. Epub 2021 Aug 31. PMID 34465915
- [Background] Tavares RM, Mendelsohn A, Grossman Y, Williams CH, Shapiro M, Trope Y, Schiller D. A Map for Social Navigation in the Human Brain. Neuron. 2015 Jul 1;87(1):231-43. doi: 10.1016/j.neuron.2015.06.011. PMID 26139376
- [Background] Constantinescu AO, O'Reilly JX, Behrens TEJ. Organizing conceptual knowledge in humans with a gridlike code. Science. 2016 Jun 17;352(6292):1464-1468. doi: 10.1126/science.aaf0941. Epub 2016 Jun 16. PMID 27313047
- [Background] Hassabis D, Kumaran D, Vann SD, Maguire EA. Patients with hippocampal amnesia cannot imagine new experiences. Proc Natl Acad Sci U S A. 2007 Jan 30;104(5):1726-31. doi: 10.1073/pnas.0610561104. Epub 2007 Jan 17. PMID 17229836
- [Background] Franklin NT, Frank MJ. Compositional clustering in task structure learning. PLoS Comput Biol. 2018 Apr 19;14(4):e1006116. doi: 10.1371/journal.pcbi.1006116. eCollection 2018 Apr. PMID 29672581
- [Background] Schuck NW, Cai MB, Wilson RC, Niv Y. Human Orbitofrontal Cortex Represents a Cognitive Map of State Space. Neuron. 2016 Sep 21;91(6):1402-1412. doi: 10.1016/j.neuron.2016.08.019. PMID 27657452
- [Background] Theves S, Fernandez G, Doeller CF. The Hippocampus Encodes Distances in Multidimensional Feature Space. Curr Biol. 2019 Apr 1;29(7):1226-1231.e3. doi: 10.1016/j.cub.2019.02.035. Epub 2019 Mar 21. PMID 30905602
- [Background] Hu X, Cheng LY, Chiu MH, Paller KA. Promoting memory consolidation during sleep: A meta-analysis of targeted memory reactivation. Psychol Bull. 2020 Mar;146(3):218-244. doi: 10.1037/bul0000223. PMID 32027149
- [Background] Yamauchi T, Markman AB. Category learning by inference and classification. Journal of Memory and language. 1998; 39(1): 124-148.
- [Background] Anderson AL, Ross BH, Chin-Parker S. A further investigation of category learning by inference. Mem Cognit. 2002 Jan;30(1):119-28. doi: 10.3758/bf03195271. PMID 11958345
- [Background] Chin-Parker S, Ross BH. The effect of category learning on sensitivity to within-category correlations. Mem Cognit. 2002 Apr;30(3):353-62. doi: 10.3758/bf03194936. PMID 12061756
- [Background] Chin-Parker S, Ross BH. Diagnosticity and prototypicality in category learning: a comparison of inference learning and classification learning. J Exp Psychol Learn Mem Cogn. 2004 Jan;30(1):216-26. doi: 10.1037/0278-7393.30.1.216. PMID 14736308
- [Background] Markman AB, Ross BH. Category use and category learning. Psychol Bull. 2003 Jul;129(4):592-613. doi: 10.1037/0033-2909.129.4.592. PMID 12848222
- [Background] Cousins JN, El-Deredy W, Parkes LM, Hennies N, Lewis PA. Cued Reactivation of Motor Learning during Sleep Leads to Overnight Changes in Functional Brain Activity and Connectivity. PLoS Biol. 2016 May 3;14(5):e1002451. doi: 10.1371/journal.pbio.1002451. eCollection 2016 May. PMID 27137944
- [Background] Cairney SA, Guttesen AAV, El Marj N, Staresina BP. Memory Consolidation Is Linked to Spindle-Mediated Information Processing during Sleep. Curr Biol. 2018 Mar 19;28(6):948-954.e4. doi: 10.1016/j.cub.2018.01.087. Epub 2018 Mar 8. PMID 29526594

RESULTS

PARTICIPANT FLOW:
Groups:
- Aim 1 Immediate Incongruent; Aim 1 Immediate Congruent: Participants will learn and be tested on two different semantic categories with the same structure that dictates the co-occurrence of different features.
  Congruent vs. Incongruent: The Congruent vs. Incongruent intervention relates to the feature-based structure of the novel categories (Modular or non-Modular) and whether there is (Congruent) or is not (Incongruent) a match between what was previously learned and the final target category.
  Immediate vs. Awake vs. Asleep: Immediate, Awake, and Sleep refer to either no break, 2.5 hours awake, or 2 hours asleep plus a 30-minute post-nap break to account for sleep inertia between learning and target category.
- Aim 2 Awake Incongruent; Aim 2 Awake Congruent: Participants will learn two different semantic categories, neither of which has a Modular structure. After a 2.5-hour break, they will learn and be tested on a novel semantic category with a Modular structure.
  Congruent vs. Incongruent: The Congruent vs. Incongruent intervention relates to the feature-based structure of the novel categories (Modular or non-Modular) and whether there is (Congruent) or is not (Incongruent) a match between what was previously learned and the final target category.
  Immediate vs. Awake vs. Asleep: Immediate, Awake, and Sleep refer to either no break, 2.5 hours awake, or 2 hours asleep plus a 30-minute post-nap break to account for sleep inertia between learning and target category.
- Aim 2 Sleep Incongruent; Aim 2 Sleep Congruent: Participants will learn two different semantic categories, one of which has a Modular structure. After a 2-hour nap opportunity, during which TMR will be used to reactivate the Modular category during rapid eye movement (REM) sleep, participants will take a 30-minute break. After the break, they will learn and be tested on a novel semantic category with a Modular structure.
  Congruent vs. Incongruent: The Congruent vs. Incongruent intervention relates to the feature-based structure of the novel categories (Modular or non-Modular) and whether there is (Congruent) or is not (Incongruent) a match between what was previously learned and the final target category.
  Immediate vs. Awake vs. Asleep: Immediate, Awake, and Sleep refer to either no break, 2.5 hours awake, or 2 hours asleep plus a 30-minute post-nap break to account for sleep inertia between learning and target category.
  Targeted memory reactivation (TMR): Targeted memory reactivation (TMR) is the systematic presentation of sounds during sleep that were associated with certain stimuli during learning and will be administered during slow wave sleep (SWS).
Period: Overall Study
Arm/Group | Aim 1 Immediate Incongruent | Aim 1 Immediate Congruent | Aim 2 Awake Incongruent | Aim 2 Awake Congruent | Aim 2 Sleep Incongruent | Aim 2 Sleep Congruent
Started | 47 | 47 | 26 | 25 | 22 | 27
Completed | 47 | 47 | 26 | 25 | 22 | 27
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Since only a small percentage of participants enter REM sleep within the 2-hour nap opportunity, if we were to randomly assign participants to either non-REM vs. REM conditions, there would be an extremely high likelihood that participants assigned to the REM condition would never enter that sleep phase, rendering that participant's data unusable and resulting in a high attrition rate. In order to generate as much usable data as possible, we therefore decided to remove the REM condition.
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Incongruent | Immediate Congruent | Awake Incongruent | Awake Congruent | Sleep Incongruent | Sleep Congruent (SWS) | Sleep Congruent (REM) | Total
Number analyzed (Participants) | 47 | 47 | 26 | 25 | 22 | 27 | 0 | 194
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
  Between 18 and 65 years | 47 | 47 | 26 | 25 | 22 | 27 |  | 194
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.0213 (1.9052) | 25.6809 (1.7706) | 21.19 (3.9) | 23.08 (4.75) | 20.95 (3.58) | 22.96 (4.42) |  | 23.67 (3.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 13 | 15 | 16 | 16 |  | 119
  Male | 17 | 18 | 13 | 10 | 6 | 11 |  | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 0 | 6 | 0 | 2 |  | 19
  Not Hispanic or Latino | 42 | 41 | 24 | 18 | 22 | 25 |  | 172
  Unknown or Not Reported | 0 | 0 | 2 | 1 | 0 | 0 |  | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 2 | 0 | 1 |  | 4
  Asian | 4 | 3 | 13 | 9 | 13 | 16 |  | 58
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
  Black or African American | 0 | 2 | 2 | 2 | 3 | 0 |  | 9
  White | 42 | 41 | 8 | 9 | 4 | 9 |  | 113
  More than one race | 0 | 1 | 1 | 1 | 1 | 1 |  | 5
  Unknown or Not Reported | 0 | 0 | 2 | 2 | 1 | 0 |  | 5
Region of Enrollment [Number; unit: participants]
  United States | 47 | 47 | 26 | 25 | 22 | 27 |  | 194

OUTCOME MEASURES:

1. Primary Outcome: Structure Knowledge for a New Modular Category in Stage 2
Description: Accuracy (0-100%) on the behavioral missing feature task in Stage 2, which requires participants to use their memory from earlier in the experiment to make a guess about how to fill in missing features of the category exemplars.
Time Frame: In Aim 1, accuracy is collected in a missing feature task 25 min. into the experiment, taking 25 min. In Aim 2, accuracy is collected in a missing feature task over 25 min in Stage 2
Measure: Mean (Standard Deviation); unit: Proportion of correct responses
Groups:
- Aim 2 Sleep Incongruent; Aim 2 Sleep Congruent: Participants will learn two different semantic categories, one of which has a Modular structure. After a 2-hour nap opportunity, during which TMR will be used to reactivate the non-Modular category, participants will take a 30-minute break. After the break, they will learn and be tested on a novel semantic category with a Modular structure.
  Congruent vs. Incongruent: The Congruent vs. Incongruent intervention relates to the feature-based structure of the novel categories (Modular or non-Modular) and whether there is (Congruent) or is not (Incongruent) a match between what was previously learned and the final target category.
  Immediate vs. Awake vs. Asleep: Immediate, Awake, and Sleep refer to either no break, 2.5 hours awake, or 2 hours asleep plus a 30-minute post-nap break to account for sleep inertia between learning and target category.
  Targeted memory reactivation (TMR): Targeted memory reactivation (TMR) is the systematic presentation of sounds during sleep that were associated with certain stimuli during learning and will be administered during slow wave sleep (SWS).
Arm/Group | Aim 1 Immediate Incongruent | Aim 1 Immediate Congruent | Aim 2 Awake Incongruent | Aim 2 Awake Congruent | Aim 2 Sleep Incongruent | Aim 2 Sleep Congruent
Number analyzed (Participants) | 47 | 47 | 26 | 25 | 22 | 27
Proportion of correct responses | 0.563 (.0983) | .5726 (.0857) | .6303 (.0942) | .6266 (.1043) | .6287 (.1147) | 0.6231 (0.0998)

ADVERSE EVENTS:
Time Frame: One day (specifically the hours during which participants were completing tasks)
Description: There were no risks in this study that could plausibly cause adverse events.
Arm/Group | Immediate Congruent | Immediate Incongruent | Awake Incongruent | Awake Congruent | Sleep Incongruent | Sleep Congruent (SWS) | Sleep Congruent (REM)
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47 | 0/26 | 0/25 | 0/22 | 0/27 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47 | 0/26 | 0/25 | 0/22 | 0/27 | 0/0
Other Adverse Events (participants affected / at risk) | 0/47 | 0/47 | 0/26 | 0/25 | 0/22 | 0/27 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT05746299/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT05746299/SAP_001.pdf
  • Informed Consent Form (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT05746299/ICF_002.pdf